CLINICAL TRIAL: NCT02925910
Title: Assesment of Patient Experience Using a Wheelchair Equipped With Suspension Wheels
Brief Title: Comparison of User Experience With Wheelsoft Wheels Intalled on a Wheelchair Compared With Normal Wheels.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 115-16emc
Record Dates: First submitted 2016-09-29; First posted 2016-10-06 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Back Pain; Personal Satisfaction; Fatigue
MeSH Terms: conditions — Back Pain; Personal Satisfaction; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- softwheels at second round (Other): Begining with regular wheelchair for 2 days and then changing for shock absorbing wheelchair for 2 days
  Interventions: Device: Shock absorbing wheelchair
- softwheels at first round (Other): starting with Shock absorbing wheelchair for 2 days and then changing for regular wheelchair for 2 days
  Interventions: Device: Shock absorbing wheelchair

INTERVENTIONS:
Device: Shock absorbing wheelchair — 2 randomised groups will try the softwheel wheelchair compare to regular one, but in different order.
  Other Names: Softwheel wheelchair

SUMMARY:
Two groups of randomised rehabilitation patients will try a softwheels wheelchair and a regular one. One group will start with the softwheelsl and then change to the regular, and the other will start with the regular and then change to the softwheel.

DETAILED DESCRIPTION:
The patients who are received to the rehabilitation ward and are confined to the use of a wheelchair are randomized to two groups. The first are given a wheelchair with wheelsoft wheels and the second group with regular wheels. The wheels of the chair are all covered to look similar to regular wheels (the regular wheels are also covered). All the patients will be taken once a day to a 10 minute trip with the wheelchair. After two days a questionnaire regarding their experience with the chair will be passed. On the third day the groups will change their wheels to the other kind. And again taken to daily trips and a final questionnaire on day four. We will collect additional data from the patients: age, sex, medical record, weight, height, ethnic background, marital status, working status.

ELIGIBILITY:
Inclusion Criteria:

* wheelchair bound for at least 4 days

Exclusion Criteria:

* not able to answer verbal questions
* over 95 kg of weight (wheel limit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-02-10 (Actual)

PRIMARY OUTCOMES:
Satisfaction - first round | 2 days
  Overall satisfaction from wheelchair (regarding pain, comfort, tiredness, muscle crumps, feeling of safety) will be measured by questionairre after the first round

SECONDARY OUTCOMES:
Satisfaction - Second round | 2 days
  Overall satisfaction from wheelchair (regarding pain, comfort, tiredness, muscle crumps, feeling of safety) will be measured by questionairre after the second round

CONTACTS AND LOCATIONS:
Overall Officials: uriel giwnewer, MD, Principal Investigator — haemek medical center
Locations (1):
- haemek MC, Afula, Israel

IPD SHARING:
Plan to Share IPD: No